CLINICAL TRIAL: NCT05709613
Title: Use of a Feedback Device to Limit Too Shallow Compressions Associated With the Use of an I-gel® Device During Simulated Out-of-Hospital Cardiac Arrest: Simulation-based Multicentre Randomised Controlled Trial
Brief Title: Use of a Feedback Device to Limit Too Shallow Compressions Associated With the Use of an I-gel® Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneve TEAM Ambulances (Other)
Responsible Party: Principal Investigator, Stuby Loric, Principal Investigator, Geneve TEAM Ambulances
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-7
Record Dates: First submitted 2023-01-08; First posted 2023-02-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Resuscitation; Emergency Medicine
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data extraction will be fully automated and the statistician will not know the identity of the participants or the sequence they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No feedback device (No Intervention): This group will have no access to the feedback device
- Feedback device (Experimental): This group will have access to the feedback device
  Interventions: Device: Use of a chest compressions' feedback device

INTERVENTIONS:
Device: Use of a chest compressions' feedback device — The participants will have access to a chest compressions' feedback device
  Arms: Feedback device

SUMMARY:
Airway management in out-of-hospital cardiac arrest is still debated. Several options exist: bag-valve-mask ventilation, supraglottic devices and endotracheal intubation. Intermediate and advanced airway management strategies could be useful devices to increase chest compression fraction. A previous study shows that early insertion of an i-gel device significantly increases chest compression fraction and enhances respiratory parameters. However, the compressions were found to be shallower in the experimental group using the i-gel device. Although, the shallower compressions found in the supraglottic airway device group did not appear to be linked to their provision in an over-the-head position, it is reasonable to assume that the addition of a feedback device to the use of an i-gel® device could fix this issue. The feedback devices seem to be able to provide a benefit, and allow deeper compressions / more often in the depth target. There is a mismatch between perceived and actual cardiopulmonary resuscitation performance supporting the need for such a feedback device's study.

ELIGIBILITY:
Inclusion Criteria:

* Registered EMTs and paramedics actively working in any of the participating study trial centers will be eligible for inclusion.

Exclusion Criteria:

* Members of the study team
* EMTs will be randomly excluded if there are more EMTs than paramedics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Compressions within the depth target | Through study completion, i.e.10 minutes of scenario.
  Proportions of compressions within the depth target of 5 to 6 centimeters

SECONDARY OUTCOMES:
Overall chest compression fraction | Through study completion, i.e.10 minutes of scenario.
  The chest compression fraction is the time during which compressions are provided divided by the total time of the resuscitation
Depth of chest compressions | Through study completion, i.e.10 minutes of scenario.
  The depth of chest compressions measured in centimeters
Compressions within the rate target | Through study completion, i.e.10 minutes of scenario.
  Proportions of compressions within the rate target of 100 to 120 compressions per minute
Rate of chest compressions | Through study completion, i.e.10 minutes of scenario.
  The rate of chest compressions measured in compressions per minute
Compressions with correct chest recoil | Through study completion, i.e.10 minutes of scenario.
  The proportions of compressions with complete chest recoil (less than 5 millimeters of deviation from the reference value)
Time to first effective ventilation | Through study completion, i.e.10 minutes of scenario.
  The time measured in seconds from beginning of the resuscitation to first effective ventilation (defined as at least 300 millilitres)

CONTACTS AND LOCATIONS:
Overall Officials: Loric Stuby, Principal Investigator — Genève TEAM Ambulances
Locations (4):
- Switzerland (4):
  - ACE Genève Ambulances, Chêne-Bougeries, Canton of Geneva
  - Ambulances de la Ville de Sion, Sion, Valais
  - Genève TEAM Ambulances, Geneva
  - SK Ambulances, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be available on Yareta as soon as the results are submitted for publication.
Supporting Information: Study Protocol
Time Frame: Once the final results will be submitted for publication
Access Criteria: Free access

REFERENCES:
- See also: Whole project website — https://swiss-cpr-studies.ch/